CLINICAL TRIAL: NCT05108285
Title: Dark Halo a New Biomarker in Macular Neovascularization: a Comparative Study Between ICGA and OCTA
Brief Title: Dark Halo and MNV: a Study Between ICGA and OCTA
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gilda Cennamo, Principal Investigator, Federico II University
Other Study IDs: 9009/21
Record Dates: First submitted 2021-10-24; First posted 2021-11-04 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Macular Neovascularisation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MNV group: Eyes affected by MNV. The dark halo of MNV was evaluated by OCTA and ICGA
  Interventions: Diagnostic Test: Optical Coherence Tomography Angiography (OCTA) and indocyanine green angiography (ICGA)

INTERVENTIONS:
Diagnostic Test: Optical Coherence Tomography Angiography (OCTA) and indocyanine green angiography (ICGA) — OCTA and ICGA is able to detect the dark halo as a area of reduced perfusion around MVN

SUMMARY:
The aim of study is to compare the evaluation of dark halo area of macular neovascularization (MNV) between indocyanine green angiography (ICGA) and optical coherence tomography angiography (OCTA) in order to identify OCTA as effective and useful biomarker in MNV

DETAILED DESCRIPTION:
Dark halo is defined as a dark perilesional of flow decrease due to an area of reduced choroidal flow adjacent to the macular neovascularization (MNV).

The detection of MNV vascular details was only possible through invasive dye injection, such as fluorescein angiography (FA) or indocyanine green angiography (ICGA).

Optical coherence tomography angiography (OCTA) is a recent imaging technique that is able to detect the perfusion and non-perfusion areas carefully.

The aim of study is to compare the evaluation of dark halo area of MNV between ICGA and OCTA

ELIGIBILITY:
Inclusion Criteria:

* age older than 55 years
* diagnosis of macular neovascularization
* absence of previous treatment with anti-Vegf injections
* absence of other retinal vascular diseases

Exclusion Criteria:

* age younger than 55 years
* absence diagnosis of macular neovascularization
* presence of previous treatment with anti-Vegf injections
* presence of other retinal vascular diseases

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A group of patients affected by MNV is subjected to OCTA and ICGA analysis in order to evaluate which of two methods is able to detect in a peculiar way the dark halo around the MNV
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Dark halo measurement | three years
  The OCTA and ICGA parameters analyzed are: the area of dark halo (mm2) that surrounds the coroidal neovascularization.

CONTACTS AND LOCATIONS:
Overall Officials: Gilda Cennamo, Principal Investigator — Università Federico II
Locations (1):
- University of Naples "Federico II", Naples, Italy

REFERENCES:
- [Derived] Fossataro F, Cennamo G, Montorio D, Clemente L, Costagliola C. Dark halo, a new biomarker in macular neovascularization: comparison between OCT angiography and ICGA-a pilot prospective study. Graefes Arch Clin Exp Ophthalmol. 2022 Oct;260(10):3205-3211. doi: 10.1007/s00417-022-05693-8. Epub 2022 May 6. PMID 35522297